CLINICAL TRIAL: NCT05046093
Title: Clinical Outcomes of Cryobiopsy for Peripheral Pulmonary Lesions - A Prospective Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2105-045-103
Record Dates: First submitted 2021-08-18; First posted 2021-09-16 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Lung Nodule
Keywords: Cryobiopsy; Pulmonary nodule; Radial EBUS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single intervention arm - transbronchial cryobiopsy (Experimental): Patients enrolled in this single arm will have lung nodules biopsied by transbronchial cryobiopsy.
  Interventions: Diagnostic Test: Transbronchial cryobiopsy

INTERVENTIONS:
Diagnostic Test: Transbronchial cryobiopsy — When the lung nodule is visualized by thin bronchoscope (4mm) with R-EBUS, cryobiopsy is performed. If not visualized, ultrathin (3mm) bronchoscope is used.
  Cryobiopsy is performed with 1.1mm cryo-probe.

SUMMARY:
As the former radial endobronchial ultrasound (R-EBUS) guided transbronchial forcep biopsy of peripheral pulmonary nodules has some limitations, the purpose of this study is to investigate a novel biopsy technique, transbronchial cryobiopsy, in patients with peripheral pulmonary nodules.

DETAILED DESCRIPTION:
This is a prospective, single arm, open label trial to assess the diagnostic accuracy and safety of the transbronchial cryobiopsy in patients with peripheral pulmonary nodule using a 1.1mm cryoprobe, combined with bronchoscope (with/without guide sheath), R-EBUS, virtual bronchoscopy navigation, and fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with peripheral lung nodule less than 30mm on CT scan referred for biopsy
* Age ≥ 18
* Written informed consent after participant's information

Exclusion Criteria:

* Central lesion (visible on bronchoscope) or presence of metastatic lymph node (not requiring radial EBUS)
* Pure GGO lesion
* Patients at increased risk of bleeding

  1. Cannot stop agents such as antiplatelet agent or anticoagulant therapy
  2. Coagulopathy: Thrombocytopenia (< 100,000/mm3) or prolonged PT (INR > 1.5)
* Patient with existing or risk of pulmonary and cardiovascular decompensation
* Intolerance to sedation
* Vulnerable groups such as pregnant woman, breast feeding, etc.
* Previously diagnosed cancer patient who needs re-biopsy for genetic susceptibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield based on pathologic diagnosis | up to 6 months
  Diagnostic yield based on pathologic diagnosis is defined as percentage of definitive pathological diagnosis by transbronchial cryobiopsy. If the bronchoscopic procedure fails to diagnose malignancy, the gold standard will be the results of additional procedures such as repeated bronchoscopic biopsy, percutaneous needle aspiration, surgical biopsy, or CT follow-up without any invasive procedure.

SECONDARY OUTCOMES:
Diagnostic yield based on clinical diagnosis | up to 6 months
  Diagnostic yield based on clinical diagnosis is defined as percentage of pathological diagnosis with suspicious results by transbronchial cryobiopsy. If the bronchoscopic procedure fails to diagnose malignancy, the gold standard will be the results of additional procedures such as repeated bronchoscopic biopsy, percutaneous needle aspiration, surgical biopsy, or CT follow-up without any invasive procedure.
Adverse events | up to 1 week
  Occurrence of bleeding, pneumothorax, and infection events (during the procedure and within 1 week after the intervention). Bleeding will be assessed as the following scale (a. mild = self-limiting bleeding, manageable with suction alone and without the need for any specific intervention; b. moderate = use of any additional intervention such as instillation of ice-cold saline or vasoconstrictive drugs, transient balloon tamponade, or therapeutic bronchoscope (external diameter 6mm); c. severe = additional prolonged monitoring or intensive care therapy after the procedure or if the bleeding was fatal). Pneumothorax will be assessed as the following scale (a. pneumothorax not requiring chest tube insertion; b. pneumothorax requiring chest tube insertion).

OTHER OUTCOMES:
Type of bronchoscope | up to 1 day
  Type of bronchoscope used is assessed as the following scale (a. thin; b. ultrathin).
Guide sheath use | up to 1 day
  Guide sheath use is assessed as the following scale (a. yes; b. no).
Radial endobronchial ultrasound probe orientation | up to 1 day
  Lesion orientation regarding radial endobronchial ultrasound probe is assessed as the following scale (a. within, concentric; b. within, eccentric; c. adjacent; d. invisible).
Procedure time in minutes and seconds | up to 1 day
  The time spent in procedure begins with the insertion of bronchoscope into vocal cord and ends with removal of bronchoscope from vocal cord.
Diameter of cryoprobe | up to 1 day
  Diameter of cryoprobe use is assessed as the following scale (a. 1.1mm; b. 1.7mm).
Number of biopsy | up to 1 day
  The number of biopsy samples is assessed.
Freezing time of cryoprobe in seconds | up to 1 day
  The freezing time of cryoprobe for sampling the lesions is assessed in seconds.
Biopsy size in millimeter | up to 1 month
  Size of biopsy tissue is assessed by pathologist for maximum and minimum diameter in millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Seop Eom, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Mok J, Kim S, Yoo WH, Jo EJ, Kim MH, Lee K, Kim KU, Park HK, Lee MK, Eom JS. Clinical outcomes of transbronchial cryobiopsy using a 1.1-mm diameter cryoprobe for peripheral lung lesions - A prospective pilot study. Respir Med. 2023 Oct;217:107338. doi: 10.1016/j.rmed.2023.107338. Epub 2023 Jun 26. PMID 37380091